CLINICAL TRIAL: NCT04716777
Title: Brief Transdiagnostic Group Cognitive-Behavioral Treatment for Adolescents With Internalizing Problems: A Randomized Waitlist Controlled Trial
Brief Title: Brief Transdiagnostic Group CBT for Adolescents With Internalizing Problems: A Randomized Waitlist Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Iceland (Other)
Collaborators: Primary Health Care Clinic, Reykjavik, Iceland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VSN-20-115
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-03

CONDITIONS: Anxiety Disorders; Depressive Disorder; Anxiety; Depression
Keywords: Transdiagnostic Cognitive-Behavioral Treatment; Cognitive-Behavioral Treatment; Group Treatment; Randomized Controlled Trial
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two conditions 8-week treatment or 8-week waitlist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Transdiagnostic GCBT (Experimental): Participants receive Brief Transdiagnostic group cognitive-behavioral treatment. Eight weekly sessions.
  Interventions: Behavioral: Brief Transdiagnostic group-based Cognitive-Behavioral Treatment
- Waitlist (No Intervention): Participants receive an 8-week waitlist condition with some attentional-control via monitoring for clinical deterioration. After a post-waitlist assessment, participants in this condition are offered the Brief Transiagnostic GCBT for eight weeks.

INTERVENTIONS:
Behavioral: Brief Transdiagnostic group-based Cognitive-Behavioral Treatment — Weekly group-based transdiagnostic CBT sessions for eight weeks.
  Arms: Brief Transdiagnostic GCBT

SUMMARY:
The investigators will evaluate a brief group-based cognitive-behavioral treatment program for adolescents aged 13-17 years with internalizing problems.

DETAILED DESCRIPTION:
Internalizing disorders (anxiety and depression) are among the most prevalent psychiatric disorders in youth. Cognitive-behavioral treatment (CBT) is well-establed treatment for internalizing disorders. The evidence originates mostly from disorder-specific CBT for youth. However, the validity of specific diagnosis has been questioned, especially because of high symptom overlap between disorders and the high rates of diagnostic comorbidity. In addition, research has suggested that depressive comorbidity is associated with reduced treatment effectiveness for primary anxiety disorder and vice versa. A recent meta-analysis, of the collective evidence of psychotherapy throught 50 years, revealed that there were no effects of disorder-specific psychotherapy for youths with one or more comorbid disorder. Which indicates that disorder-specific treatment is not sufficient for children with comorbidity.

Transdiagnostic treatments have been developed and evaluated to address this problem. These treatments emphasize effective therapeutic principles which may be applied across multiple disorders. Transidagnostic treatment may be more cost effective and practical than disorder-specific treatments as most therapists only need to be trained extensively in one protocol. Transdiagnostic treatments may also be easily learned by clinicians and especially in generalist settings where one transdiagnostic protocol can be offered to patients with various mental health problems instead of many offered to much fewer. Offering transdiagnostic treatment approach may better serve the diagnostically heterogeneous groups which seek help at general clinics instead of many different disorder-specific treatment protocols. Transdiagnostic CBT protocols have been proved to be effective among adults with internalizing disorders and also among youths. It has also been showed that transdiagnostic CBT was equally effective as anxiety disorder-specific protocol for adults with anxiety disorders.

Treatment Our treatment is a brief group-based cognitive-behavioral treatment which was specifically designed for adolescents with impairing internalizing symptoms, or anxiety/depressive disorders seeking help at the Primary Health Care Clinics in Iceland. The treatment comprises eight weekly 110-minutes sessions were the following components are applied: (1) psychoeducation, (2) cognitive restructuring, (3), behavioral activation, (4) exposure, (5) problem solving, (6) social skills, and (7) mindfulness. The participants receive a workbook with outline of each sessions and assignments related to components (e.g., (e.g., ABC workseets, exposure exercises). They are encouraged to practice skills learned in sessions between sessions. All parents attend two sessions. They receive detailed psychoeducation and are instructed in assisting their children with the homework assignments (week 1), and in week 6 they are instructed how to assist their children with exposure exercises. They also receive a workbook with outline of each sessions. The therapist also has at least one telephone call with each family to follow-up on exercises.

Study design and participants The following study is a randomized controlled trial where participants are allocated to either eight weekly sessions of brief transidagnostic CBT or waitlist monitoring for clinical deterioration. The investigators will randomize by using blockwise procedure determined by a computer-generated algorithm. To ensure that the randomization will not be predicted in advance, it will be centralized at the University of Iceland. Participants will be assigned to study group after being deemed eligible and undergoing consent.

Assessment Participants will be assessed at baseline, midtreatment, posttreatment (week 8), 2 months follow-up, 4 months follow-up, and 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1 SD above normal population mean on the Revised Children's Anxiety and Depression Scale (parent- or self-report), subscale or total score OR a K-SADS-PL confirmed anxiety or depressive disorder.

Exclusion Criteria:

* Inadequate language proficiency by the patient or the parent.
* The presence of other psychiatric disorders having a higher treatment priority (i.e., psychosis and acute sucide risk)
* Intellectual Disability

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Revised Children's Anxiety and Depression Scale (RCADS) | Measured at baseline, week 4, and week 8 (post-treatment). Measured at 2-, 4-months, and 1-year follow-up (open trial)
  Self-report total score of anxiety / depression

SECONDARY OUTCOMES:
Parent-report of the Revised Children's Anxiety and Depression Scale (RCADS) | Measured at baseline, week 4, and week 8 (post-treatment). Measured at 2-, 4-months, and 1-year follow-up (open trial)
  Parent-report total score of anxiety / depression
KINDL Quality of life, parent- and self-report | Measured at baseline and week 8 (post-treatment). Measured at 2-, 4-months, and 1-year follow-up (open trial)
  generic instrument for assessing Health-Related Quality of Life in children and adolescents
Clinical reliable change and clinical significant change | Measured at baseline, week 4, and week 8 (post-treatment). Measured at 2-, 4-months, and 1-year follow-up (open trial)
  Based on the RCADS self-report using the approach by Jacobson and Truax

CONTACTS AND LOCATIONS:
Overall Officials: Gudmundur Skarphedinsson, PhD, Principal Investigator — University of Iceland
Locations (1):
- Primary Health Care Clinic, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No